CLINICAL TRIAL: NCT05428449
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of GT20029 Following Topical Single and Multiple Ascending Dose Administration
Brief Title: Study in Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of GT20029
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT20029-US-1001
Record Dates: First submitted 2022-03-15; First posted 2022-06-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Androgenetic Alopecia; Acne Vulgaris
MeSH Terms: conditions — Alopecia; Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GT20029 (Experimental)
  Interventions: Drug: GT20029 Gel
- GT20029 Placebo (Placebo Comparator)
  Interventions: Drug: GT20029 Gel Placebo

INTERVENTIONS:
Drug: GT20029 Gel — Stage 1: One single dose Stage 2: One single dose per day (QD) or twice a day (BID) treatment over 14-day period
  Arms: GT20029
Drug: GT20029 Gel Placebo — Stage 1: One single dose Stage 2: One single dose per day (QD) or twice a day (BID) treatment over 14-day period
  Arms: GT20029 Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel group, dose escalation study to evaluate the safety, tolerability and pharmacokinetics (PK) of GT20029 following topical single ascending dose in healthy subjects and multiple ascending dose administration in subjects with androgenetic alopecia(AGA) or acne

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria can be enrolled into the study:

  1. For all(Cohort 1+ 2):

     1. Aged 18 to 60 years old;
     2. The subject or legally authorized representative gives signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol;
     3. Understand and agree to comply with planned study procedures;
     4. Subjects with a weight of ≥ 50 kg for male, a weight of ≥ 45 kg for female, and a body mass index (BMI) between 19 and 30 kg/m2 (inclusive);
     5. Subjects are able to communicate well with the investigator and understand and comply with the requirements of the study
     6. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs.
  2. For Cohort 1(single dose escalation):

     1. Healthy subjects, male or non-pregnant female;
     2. The subject's skin is healthy without damage or wound, tattoos and scars;
  3. For Cohort 2a(multiple dose escalation):

     1. Male;
     2. Have a clinical diagnosis of mild to moderate androgenetic alopecia; rating IIIv, IV and V on the modified Norwood Hamilton Scale, with a history of ongoing hair loss；
     3. Subject is willing to maintain the same hairstyle, hair length, and hair color throughout the study；
  4. For cohort 2b (multiple dose escalation)

     1. Male or non-pregnant female;
     2. Subjects clinically diagnosed with grade I-III acne vulgaris as per the Pillsbury International Modified Classification, and with an IGA score of 2-3;
     3. Subject has used the same type and brand of make-up, other facial products (exclusive of RX/OTC acne cleansers) and hair products (e.g., shampoo, gel, hair spray, mousse, etc.) for at least one (1) month prior to the Baseline Visit and agrees to continue his/her other general skin and hair care products and regimen for the entire study.
  5. Negative COVID-19 results within 7 days prior first dosing

Exclusion Criteria:

* Subjects will be excluded from study entry if any of the following exclusion criteria are present at screening:

  1. For all:

     1. Prior allergy to the investigational drug or any components;
     2. Use of drugs with the same target and mechanism as the investigational drug (androgen receptor degradation agent) within 1 month prior to screening;
     3. Any visible skin disease, damage or condition at the application site which, in the opinion of the investigator, could compromise subject safety and/or interfere with the evaluation of the test site reaction;
     4. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity
     5. Known or suspected malignancy;
     6. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
     7. A hospital admission or major surgery within 30 days prior to screening;
     8. Participation in any other investigational drug trial within 30 days prior to screening;
     9. A history of drug abuse within 6 months prior to screening or a positive screen for drugs of abuse;
     10. Subjects with an alcohol consumption of more than 14 units per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to signing the informed consent form, or subjects with a positive breath alcohol test result the day before dosing (breath alcohol content > 0.0 mg/100 mL), or subjects cannot abstain from alcohol during the study;
     11. Subjects with a previous chronic consumption of excessive (more than 8 cups a day, 1 cup = 200 mL) tea, coffee, or caffeine-containing beverages;
     12. Subjects with a consumption of any food or beverages containing caffeine, alcohol, xanthine or grapefruit (e.g., coffee, strong tea, chocolate, etc.) within 48 hours prior to the first dose;
     13. Subjects who have difficulty in blood collection or cannot tolerate venipuncture or have a history of fear of needles and hemophobia;
     14. Subjects with a blood donation history or blood loss of ≥ 200 mL within 3 months prior to the study, or who plan to donate blood or blood components during the study or within 3 months after the end of the study;
     15. Subjects who smoked more than 5 cigarettes per day within 3 months before the study and who could not stop smoking during the entire study;
     16. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
     17. Use of prescription or over-the-counter (OTC) medications, and herbal (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing);
     18. An unwillingness to use highly effective contraceptive measures if engaging in sexual intercourse with a partner of childbearing potential. Highly effective measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone subdermal implants, or a tubal ligation, and men or women who are unwilling to use contraception throughout the study and until 1 month after the end of the study.
     19. Subjects who are employees or related personnel of the investigator, study site, sponsor, and contract research organization;
     20. Subjects who have other conditions that may affect compliance in the opinion of the investigator, or who are unable to participate in the study for his/her own reasons;
     21. Subjects who are unable to communicate or cooperate with health care professional due to neurological, psychiatric or language disorders
  2. For Cohort 2a (subjects with alopecia):

     1. Subject has any dermatological disorders of the scalp in the target region with the possibility of interfering with the application of the investigational drug, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy;
     2. Subject has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the investigational drug or requires use of interfering topical, systemic (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns), or surgical therapy;
     3. Subject has current or recent history (within 12 months) of hair weaves, non-breathable wigs, or hair bonding;
     4. Subject had scalp hair transplants at any time;
     5. Subject has a history or active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania, or conditions/diseases other than AGA;
     6. Subject has a current or recent history (within six months) of severe dietary or weight changes or has a history of eating disorder(s); if such has resulted in hair loss refer to exclusion criterion #5;
     7. Any disorder, including but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could affect the safety of the subject throughout the study
  3. For Cohort 2b(acne)

     1. Subject has greater than two (2) facial nodules.
     2. Subject has nodulocystic acne.
     3. Subject has facial hair that could interfere with the study assessments in the opinion of the investigator.
     4. Subject has used any of the following topical anti-acne preparations or procedures on the face:

        * Topical anti-acne treatments including, but not limited to, over-the-counter (OTC) acne cleansers or treatments, benzoyl peroxide, antibiotics, azelaic acid, sulfa based products, corticosteroids and salicylic acid within two (2) weeks of the initiation of treatment.
        * Retinoids, including tazarotene, adapalene, tretinoin, within four (4) weeks of the initiation of treatment.
        * Light treatments, microdermabrasion, or chemical peels within eight (8) weeks of the initiation of treatment.
     5. Subject has used the following systemic anti-acne medications:

        * Corticosteroids (including intramuscular and intralesional injections) within four (4) weeks of the initiation of treatment. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable (stable use is defined as dose and frequency unchanged for at least four (4) weeks prior to the initiation of treatment).
        * Antibiotics within four (4) weeks of the initiation of treatment with the exception of five (5) days or less of antibiotic therapy during this period, BUT with no antibiotics use permitted within one (1) week prior to the initiation of treatment.
        * Spironolactone within eight (8) weeks of the initiation of treatment with the exception of five (5) days or less of spironolactone therapy during this period, BUT with no spironolactone use permitted within one (1) week prior to the initiation of treatment.
        * Retinoid therapy within six (6) months of the initiation of treatment.
        * Other systemic therapy which may materially affect the subject's acne in the opinion of the investigator.
  4. For female subjects:

     1. Pregnant, lactating women, or women who plan to become pregnant during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Adverse event | Stage 1 is about 22 days and stage 2 is about 35 days
  8 subjects in a group do not experience any Grade 3 or higher AEs (assessed by NAIDS 2017 v2.1) within 7 days after the last dose, the dose can be escalated to the next.
  Dose-escalation will be stopped if any of the following occur:
  * a SAE occurs in one or more active-treated subjects that is considered probably or definitely related to study drug
  * ≥50% subjects receiving active treatment experience a severe non-serious adverse event that is considered probably or definitely related to study drug
  * ≥50% subjects receiving active treatment experience, for example, a Grade 2 or higher cardiac or bone marrow adverse event or Grade 3 or higher adverse event for other systems
Skin irritation assessments | Stage 1 is about 22 days and stage 2 is about 35 days
  Dose-escalation will be stopped if any of the following occur:
  • ≥2 subjects receiving active treatment in a group experience one (or more) severe local skin reaction (score = 5, 6 or 7)
To characterize the PK Cmax of GT20029 | Stage 1 is about 22 days and stage 2 is about 35 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1 and 2: Cmax
To characterize the PK Tmax of GT20029 | Stage 1 is about 22 days and stage 2 is about 35 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1 and 2: Tmax
To characterize the PK t1/2 of GT20029 | Stage 1 is about 22 days and stage 2 is about 35 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is Stage 1: t1/2
To characterize the PK AUC of GT20029 | Stage 1 is about 22 days and stage 2 is about 35 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1 and Stage 2: AUC

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Velocity San Diego, San Diego, California
  - JBR Clinical Research Sharp, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No